CLINICAL TRIAL: NCT02989363
Title: Evaluation of the Use of Resources and Costs With O-arm in Brain Stimulation Deep Surgeries and Complex Back Surgeries
Brief Title: Evaluation of the Use of Resources and Costs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Study ECOPRES
Record Dates: First submitted 2016-11-29; First posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-11

CONDITIONS: Surgical Incision
Keywords: deep brain surgery and complex back surgery
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- O-Arm in deep brain stimulation surgeries (DBS) (Experimental): Use of image surgery with technology O-Arm in deep brain stimulation surgeries (DBS)
  Interventions: Procedure: Device O-Arm in DBS
- Control group Not O-Arm in deep brain stimulation surgeries (Experimental): Not use of image surgery with technology O-Arm in deep brain stimulation surgeries (DBS)
  Interventions: Procedure: Not device O-Arm in DBS
- O-Arm in complex back surgeries (RAQUIS) (Experimental): Use of image surgery with technology O-Arm in complex back surgeries (RAQUIS)
  Interventions: Procedure: Device O-Arm in RAQUIS
- Control group Not O-Arm in complex back surgeries (RAQUIS) (Experimental): Not use of image surgery with technology O-Arm in complex back surgeries (RAQUIS)
  Interventions: Procedure: Not device O-Arm in RAQUIS

INTERVENTIONS:
Procedure: Device O-Arm in DBS — Deep brain stimulation surgeries with device O-Arm
  Arms: O-Arm in deep brain stimulation surgeries (DBS)
Procedure: Device O-Arm in RAQUIS — Complex back surgeries with the device O-Arm
  Arms: O-Arm in complex back surgeries (RAQUIS)
Procedure: Not device O-Arm in DBS — Deep brain stimulation surgeries without the device O-Arm
  Arms: Control group Not O-Arm in deep brain stimulation surgeries
Procedure: Not device O-Arm in RAQUIS — Complex back surgeries without the device O-Arm
  Arms: Control group Not O-Arm in complex back surgeries (RAQUIS)

SUMMARY:
Evaluation of the use of resources and costs with O-arm in deep brain stimulation (DBS) surgeries and complex back surgeries

DETAILED DESCRIPTION:
To measure the use of health resources in application A (with DBS) and in application B (vertebral fusions), in patients in the intervention group with O-arm and in the control group (usual care without O-arm) with the cost in each phase (pre-surgical, surgical, post-surgical and follow-up at 6 months (RAQUIS) and at 12 months (DBS))

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years.
* Signed informed consent.
* Patients with indication for DBS surgery for movement disorders, epilepsy and obsessive-compulsive disorder, or for cervical, dorsal or lumbar fusion surgery levels 1,2 and 3 in a degenerative disease

Exclusion Criteria:

* Patients who have had pediatric instrumented surgery.
* Patients in which the pedicle screws are inserted for neoplasia or other disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Costs of health resources (stays, visits, diagnostic and therapeutic tests, personnel, consumables and implants) with DBS (O-Arm and without O-Arm groups) | 12 months
Costs of health resources (stays, visits, diagnostic and therapeutic tests, personnel, consumables and implants) with vertebral fusions (O-Arm and without O-Arm groups) | 6 months

SECONDARY OUTCOMES:
Safety of surgeries in the control group (RAQUIS) measured like rate of complications associated with surgery | 6 months
Safety of surgeries in the intervention groups (DBS) measured like rate of complications associated with surgery | 12 months
Quality of life related to health in the intervention group (DBS) measured with the EQ-5D questionary | 12 months
Accuracy of surgeries in the control group (RAQUIS) measured with the rate of electrode or thyroid replacement during surgery | 6 months
Accuracy of surgeries in the intervention group (DBS) measured with the rate of electrode or thyroid replacement during surgery | 12 months
Safety of surgeries in the control group (RAQUIS) measured like rate rate of surgical re-intervention | 6 months
Safety of surgeries in the intervention groups (DBS) measured like rate of surgical re-intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Botella, Principal Investigator — Instituto de Investigación Sanitaria La Fe
Locations (1):
- Instituto de Investigación Sanitaria La Fe, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided